CLINICAL TRIAL: NCT06947070
Title: "Comparative Evaluation of Surface Topography and Color Stability of Implant Supported Provisional Restorations Fabricated Using Two Different 3D Printing Materials in Mandibular Posterior Region: A Randomized Clinical Trial"
Brief Title: Surface Topography and Color Stability of Implant Supported 3D Printed Provisional Restorations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Dr. Kritika Diwan
Record Dates: First submitted 2024-06-13; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: DENTAL IMPLANTATION
Keywords: 3D printed provisional restorations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- To evaluate the surface topography and color stability of Group I 3D printing provisional material. (Active Comparator)
  Interventions: Procedure: To evaluate the surface topography and color stability of 3D printing provisional material.
- To evaluate the surface topography and color stability of Group II 3D printing provisional material. (Active Comparator)
  Interventions: Procedure: To evaluate the surface topography and color stability of 3D printing provisional material.

INTERVENTIONS:
Procedure: To evaluate the surface topography and color stability of 3D printing provisional material. — Subjects with single stage implant placement followed by early non-functional loading with implant supported provisional restorations fabricated using 3D printing provisional material.

SUMMARY:
Patient attending the Outdoor Patient Department of the Department of Prosthodontics at Post Graduate Institute of Dental Sciences, Rohtak will be screened. The screening will include history taking and clinical examination of the partially edentulous patients. Patients will be selected according to the inclusion and exclusion criteria. Single stage endosseous implants will be placed. Two different Biocompatible 3D printed Polymethyl methacrylate resin will constitute two groups, Group A and Group B. 3D printed provisional poly methyl methacrylate resin crowns will be fabricated with Group- A and Group-B material followed by evaluation of surface topography and color stability after intraoral use.

DETAILED DESCRIPTION:
Title: "Comparative Evaluation of Surface Topography and Color Stability of Implant Supported Provisional Restorations Fabricated using Two Different 3D Printing Materials in Mandibular Posterior Region: A Randomized Clinical Trial".

Rationale: The study needs to verify the surface topography and color stability of implant supported provisional restorations fabricated using two different 3D printing materials in mandibular posterior region.

Aim and objectives: To evaluate the surface topography and color stability of implant supported provisional restorations fabricated using two different 3D printing materials in mandibular posterior region.

Setting: Department of Prosthodontics and Crown & Bridge, PGIDS Rohtak. Study Design: Randomised clinical trial. Population/Participants: Provisional restoration will be fabricated using two different 3D printing materials.

Sample Size: Total of 24 samples will be prepared (n=12 samples per test group).

Methodology: This is an in-vivo study and will be carried out in the Department of Prosthodontics and Crown & Bridge, Post Graduate Institute of Dental Sciences, Rohtak with the purpose to evaluate the surface topography and color stability of implant supported provisional restorations fabricated using two different 3D printing materials in mandibular posterior region.

Outcome Measures: Measuring the surface topography using profilometer and color stability using spectrophotometer.

Statistical Analysis: Data obtained would be compiled on MS Office Excel Sheet (v 2010) and will be subjected to statistical analysis using statistical package for social sciences (SPSS v 21.0, IBM). Intergroup and intragroup comparisons will be done according to distribution of data.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects consented to participate in the study.
2. Subjects with maintainable oral hygiene.
3. Subjects with adequate edentulous space at the prospective implant site.
4. Subjects with availability of adequate quantity and quality of bone.

Exclusion Criteria:

1. Subject with presence of infection around proposed site of implant placement.
2. Subjects with any condition that would interfere with the soft tissue and bone healing.
3. Subjects in which surgical procedure is contraindicated for any reasons.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-04-24 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Surface topography of provisional restorations. | 2 years
  The surface topography of implant supported provisional restorations fabricated using two different 3D printing materials evaluated using Profilometer.
Color stability of provisional restorations | 2 years
  The color stability of implant supported provisional restorations fabricated using two different 3D printing materials evaluated using Spectrophotometer.

CONTACTS AND LOCATIONS:
Overall Officials: Kritika Diwan, BDS, Principal Investigator — PGIDS, Rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No